CLINICAL TRIAL: NCT00261716
Title: Motivational Interviewing to Improve Work Outcomes in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: O3176-R
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-06

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: clinical trial; employment; schizoaffective disorder; schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPS and VOMI (Experimental): Individual Placement and Support (IPS), a form of evidence-based supported employment with 4 sessions of manualized vocationally-oriented motivational interviewing (VOMI) prior to each course of job searching
  Interventions: Behavioral: IPS; Behavioral: VOMI
- IPS and IE (Active Comparator): Individual placement and support (IPS), a form of evidence-based supported employment with 4 sessions of education about schizophrenia/schizoaffective disorder (IE), as appropriate, prior to each course of job searching
  Interventions: Behavioral: IPS; Behavioral: IE

INTERVENTIONS:
Behavioral: IPS — Individual Placement and Support Evidence based supported employment
Behavioral: IE — Four sessions of manualized illness education about schizophrenia/schizoaffective disorder (tailored to the participant diagnosis) prior to each course of a job search
  Arms: IPS and IE
Behavioral: VOMI — Four sessions of manualized motivational interviewing oriented to employment goals and concerns prior to each course of a job search
  Arms: IPS and VOMI

SUMMARY:
Many persons with schizophrenia have difficulty getting and keeping a job. This study is designed to compare the benefits of four sessions of motivational interviewing or illness education in increasing employment rates accruing from participation in supported employment.

DETAILED DESCRIPTION:
Many individuals with serious psychiatric illnesses wish to work, and yet employment rates for this population are lower than the general population (Cook & Razanno, 2000). IPS is a type of supported employment intervention designed to assist individuals with serious psychiatric illnesses return to work. Over 20 randomized trials demonstrate that, in comparison to control conditions such as group therapy or referrals to traditional vocational rehabilitation services, IPS participants are three more times more likely to obtain a job during the study, and at least twice as likely to be competitively employed at any point in the study. Just as with the general population, the rewards of work for individuals with serious mental illness include considerably more than the financial remuneration. For example, employment appears to confer higher self-esteem, greater life satisfaction, and perhaps even better treatment compliance, symptom improvement, and insight in persons with psychiatric illnesses (Bell et al, 1996; Lysacker et al, 1995; Mueser et al, 1997; Bond et al, 1997; Kashner et al, 2002). Despite its demonstrated effectiveness, these IPS results could be improved. Most IPS participants are not competitively employed at any point in time, it takes an average of about four months to obtain a first job, a typical job lasts only approximately 20-25 weeks, and employment rates across the sample asymptote at about month 8 or 9 of participation in the trials. Furthermore, obtaining a first job seems to be an almost insurmountable impediment for approximately 35-40% of individuals in the trials, and these findings may be worse in individuals iwth schizophrenia (Twamely et al, 2003) . Motivational deficits may play a prominent role in explaining the limited benefits accruing from IPS in persons with serious and persisting psychiatric illnesses, especially in those with schizophrenia. Building a successful work life requires sustained effort over months and years (Palmer, 1989). After a period of unemployment, individuals must obtain their first reemployment position, and then transition to others as circumstances arise. Many persons with schizophrenia experience high degrees of negative symptoms, demoralization, and ambivalence, which likely all interfere with the persistent efforts required to initiate and maintain a successful vocational adjustment. Enhancing already validated vocational rehabilitation programs, such as IPS, with specific techniques to address motivational deficits may be essential to increasing employment rates among persons with schizophrenia. In this study, we tested a novel strategy designed to improve motivation for positive behavior change, motivational interviewing, adapted for work-related problems, in persons with schizophrenia. With the objective of improving work outcomes, we assigned 38 outpatients with schizophrenia or schizoaffective disorder to one of two 18 month psychosocial treatment groups, traditional Individual Placement and Support (IPS) with the addition of illness education (IE) about schizophrenia/schizoaffective disorder, as appropriate, or with the addition of Vocationally-oriented Motivational Interviewing (VOMI). We hypothesized that: 1) clients with schizophrenia who participated in IPS+VOMI would better vocational outcomes than IPS+IE clients. 2) If they are separated from their first job, clients with schizophrenia who participate in IPS+VOMI would be more likely to obtain a second job than clients who receive IPS+IE; and 3) Regardless of their treatment condition, working clients with schizophrenia would have greater social adjustment, symptoms, and life satisfaction than those who are not working.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have schizophrenia or schizoaffective disease
* Currently unemployed but want to get at least a part time job
* Be on a stable medication regimen and compliant with treatment
* Live within one hour of the hospital
* Be willing to have care transferred to the Schizophrenia Outpatient Clinic at VA Greater Los Angeles Healthcare System

Exclusion Criteria:

* Organic brain disease
* Physical illnesses that would preclude working

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley M. Glynn, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI for access to data

RESULTS

PARTICIPANT FLOW:
Groups:
- IPS+VOMI: Individual Placement and Support (IPS), a form of evidence-based supported employment with 4 sessions of manualized vocationally-oriented motivational interviewing (VOMI) prior to each course of job searching
  Individual Placement and Support (IPS): Evidence based supported employment
  Vocationally-Oriented Motivational Interviewing (VOMI): Four sessions of manualized motivational interviewing oriented to employment goals and concerns prior to each course of a job search
- IPS+IE: Individual placement and support (IPS), a form of evidence-based supported employment with 4 sessions of education about schizophrenia/schizoaffective disorder (IE), as appropriate, prior to each course of job searching
  Individual Placement and Support (IPS): Evidence based supported employment
  Illness Education (IE): Four sessions of manualized illness education about schizophrenia/schizoaffective disorder (tailored to the participant diagnosis) prior to each course of a job search
Period: Overall Study
Arm/Group | IPS+VOMI | IPS+IE
Started | 17 | 21
Completed | 11 | 11
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPS+VOMI | IPS+IE | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.94 (11.08) | 40.71 (12.72) | 41.26 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 11 | 19 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8 | 7 | 15
  African American | 6 | 8 | 14
  Asian | 1 | 3 | 4
  Hispanic | 2 | 2 | 4
  Other | 0 | 1 | 1
Education [Number; unit: participants]
  12 years or less | 5 | 9 | 14
  Some College | 8 | 10 | 18
  College Graduate | 3 | 2 | 5
  missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Obtained Employment
Description: Number of participants who obtained a competitive job
Time Frame: 18 months of study
Measure: Number; unit: participants
Arm/Group | IPS+VOMI | IPS+IE
Number analyzed (Participants) | 17 | 21
participants
  Obtained at least one job | 7 | 12
  Never worked | 10 | 9
Statistical Analysis 1: Comparison: IPS+VOMI vs IPS+IE; Intent to treat analysis; Test type: Superiority or Other; p = .33, Chi-squared; 1 degree of freedom

2. Primary Outcome: Average Number of Days Worked
Description: Average number of total days each participant worked in the study
Time Frame: 18 months of study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IPS+VOMI | IPS+IE
Number analyzed (Participants) | 17 | 21
days | 93.47 (163.7) | 110 (147.8)
Statistical Analysis 1: Comparison: IPS+VOMI vs IPS+IE; intent to treat analysis; Test type: Superiority or Other; p = .75, t-test, 2 sided; degrees of freedom=36

3. Primary Outcome: Average Number of Hours Worked Per Week For Those Who Worked
Description: Average number of hours worked per week among participants who obtained a job
Time Frame: 18 months of study
Population: Only included hours worked for participants who obtained a job (n=19 in the entire study)
Measure: Mean (Standard Deviation); unit: hours/worked per week
Arm/Group | IPS+VOMI | IPS+IE
Number analyzed (Participants) | 7 | 12
hours/worked per week | 18.24 (13.77) | 13.10 (12.24)
Statistical Analysis 1: Comparison: IPS+VOMI vs IPS+IE; Test type: Superiority or Other; p = .41, t-test, 2 sided; degrees of freedom=17

4. Secondary Outcome: Obtained a Second Job if Lost First Job and Still Had at Least 2 Months in the Program
Description: Number of participants who obtained a second or third job if lost his/her first job but still had at least 2 months in the study
Time Frame: 18 months of the study
Population: Includes only participants who obtained at least one job and had at least 2 months left if they lost/left that job; 2 individuals in each condition held the same job for almost the whole program and thus could not contribute data here
Measure: Number; unit: participants
Arm/Group | IPS and VOMI | IPS and IE
Number analyzed (Participants) | 5 | 10
participants
  Held one job | 3 | 8
  Held more than one job | 2 | 2
Statistical Analysis 1: Comparison: IPS and VOMI vs IPS and IE; intent to treat --all participants who obtained at least one job; Test type: Superiority or Other; p > .05, Fisher Exact; Fishers exact= 1.0; one degree of freedom
Statistical Analysis 2: Comparison: IPS and VOMI vs IPS and IE; Test type: Superiority or Other; p > .05, Fisher Exact

5. Secondary Outcome: Association Between Employment Status and Psychiatric Symptoms as Measured on the Brief Psychiatric Rating Scale
Description: Employment status at each major follow-up assessment period and psychiatric symptomatology as reflected in the Total Brief Psychiatric Rating Scale Score (Ventura J, et al., Training and quality assurance with the Structured Clinical Interview for DSM-IV (SCID-I/P). Psychiatry Research, 1998. 79(2): p. 163-173) with scale range from 24 to 168, with higher scores indicating greater symptomatology
Time Frame: 6,12, 18 months
Population: Number of individuals working within one month of assessment point varies by follow up point; total n=38 at baseline; total n=23 analyzed at 6 months; total n= 19 analyzed at 12 months; total n = 16 analyzed at 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Employed: Participant indicated he/she was employed at least part-time within one month of scheduled assessment
- Not Employed: Participant indicated he/she was not employed at least part-time within one month of scheduled assessment
Arm/Group | Employed | Not Employed
Number analyzed (Participants) | 19 | 19
units on a scale
  6 month | 39.88 (7.40) | 42.20 (7.77)
  12 months | 41.17 (5.49) | 41.92 (8.69)
  18 months | 39.63 (5.83) | 37.75 (3.54)
Statistical Analysis 1: Comparison: Employed vs Not Employed; Intent to treat analysis; Test type: Superiority or Other; p = .37, Mixed Models Analysis; employment status effect- F(1,12)=..85
Statistical Analysis 2: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .16, Mixed Models Analysis; time effect F(1,54)=.2.05
Statistical Analysis 3: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .63, Mixed Models Analysis; employment status X time effect F (1,54)=.. 24

6. Secondary Outcome: Association Between Employment Status and Self-reported Life Satisfaction Measured on the Quality of Life Scale (Lehman)
Description: Employment status at each major follow-up assessment period and self-reported Life Satisfaction (range from 1 (terrible) to 7 (delighted)) on the Quality of Life Scale (Lehman A, Kernan E, and Postrado L, Toolkit for Evaluating Quality of Life for Persons with Severe Mental Illness. 1995, Baltimore, MD: The Evaluation Center at HSRI).
Time Frame: 6,12, 18 months
Population: Number of individuals working within one month of assessment point varies by follow up point; total n=38 at baseline; total n=26 analyzed at 6 months; total n= 19 analyzed at 12 months; total n = 17 analyzed at 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Employed | Not Employed
Number analyzed (Participants) | 19 | 19
units on a scale
  6 month | 5.00 (1.07) | 5.11 (1.08)
  12 months | 5.50 (1.05) | 4.69 (1.44)
  18 months | 5.0 (.93) | 5.44 (.53)
Statistical Analysis 1: Comparison: Employed vs Not Employed; intent to treat analysis; Test type: Superiority or Other; p = .62, Mixed Models Analysis; employment status effect F(1,12)=.26
Statistical Analysis 2: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .65, Mixed Models Analysis; time effect F (1,58)=.21 ,
Statistical Analysis 3: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .81, Mixed Models Analysis; employment status X time effect F(1,58)=.06

7. Secondary Outcome: Association Between Employment Status and Overall Adjustment as Rated on the Social Adjustment Scale II (Schooler)
Description: Employment status at each major follow-up assessment period and overall adjustment as rated on the Social Adjustment Scale II (Schooler, N., G. Hogarty, and M. Weissman, Social Adjustment Scale II (SAS-II), in Resource Materials for Community Mental Health Program Evaluations, W.A. Hargreaves, C.C. Atkisson, and J.E. Sorenson, Editors. 1979, NIMH: Rockville, MD. p. 290-303), on a 1 (excellent adjustment ) to 7 (severe maladjustment) scale.
Time Frame: 6, 12, and 18 months
Population: Number of individuals working within one month of assessment point varies by follow up point; total n=38 at baseline; total n=25 analyzed at 6 months; total n= 16 analyzed at 12 months; total n = 17 analyzed at 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Employed | Not Employed
Number analyzed (Participants) | 19 | 19
units on a scale
  6 month | 3.63 (.52) | 4.29 (.77)
  12 months | 3.75 (.50) | 4.17 (.72)
  18 months | 3.13 (.35) | 4.0 (1.0)
Statistical Analysis 1: Comparison: Employed vs Not Employed; Intent to treat analysis; Test type: Superiority or Other; p = .19, Mixed Models Analysis; employment status effect F(1,12)=1.95,
Statistical Analysis 2: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .09, Mixed Models Analysis; time effect (1.54)=2.99,
Statistical Analysis 3: Comparison: Employed vs Not Employed; Test type: Superiority or Other; p = .39, Mixed Models Analysis; employment status X time effect (F(1,54)=.74

ADVERSE EVENTS:
Time Frame: Length of Study--18 months
Description: Information obtained from routine medical chart review and every 6 month interviews with participants
Arm/Group | IPS+VOMI | IPS+IE
Serious Adverse Events (participants affected / at risk) | 6/17 | 5/21
Other Adverse Events (participants affected / at risk) | 1/17 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPS+VOMI (N=17) | IPS+IE (N=21)
Hospitalization or ER visit (Psychiatric disorders) | 6 (7) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPS+VOMI (N=17) | IPS+IE (N=21)
Torn tendon in finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Increased psychiatric symptoms (Psychiatric disorders) | 0 (0) | 3 (3) — Anxiety depression, or suspiciousness,
Elevated blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leg infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size reflecting recruitment challenges

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes